CLINICAL TRIAL: NCT03535051
Title: The Efficiency of Fractional-Laser Resurfacing Followed by Topical Tacrolimus 0.03% Cream Versus Topical Tacrolimus Alone in Stable Vitiligo: a Comparative Study
Brief Title: Efficiency of Fractional-Laser Resurfacing Followed by Topical Tacrolimus 0.03% Cream vs Tacrolimus Alone in Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Nuhah Omar, Resident, Kasr El Aini Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2018-05-12; First posted 2018-05-24 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Stable Vitiligo
Keywords: vitiligo; fractional carbon dioxide laser; tacrolimus; drug delivery
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: A total of 152 lesions in different areas of the body were evaluated in the study. Seventy six lesions received the combination treatment and 76 received topical tacrolimus alone. Forty six lesions were in the head and neck region, 40 were acral in location, 36 were in the upper and lower limbs, 22 lesions were over bony prominences and 8 lesions were present on the trunk.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (Experimental): Combination treatment of fractional carbon dioxide laser monthly sessions and topical tacrolimus 0.03% daily application (Tacrolimus Oint 0.03%)
  Interventions: Device: fractional carbon dioxide laser; Drug: Tacrolimus Oint 0.03%
- Treatment B (Active Comparator): Monotherapy with only topical tacrolimus 0.03% daily intervention: Tacrolimus Oint 0.03%
  Interventions: Drug: Tacrolimus Oint 0.03%

INTERVENTIONS:
Device: fractional carbon dioxide laser — Monthly fractional carbon dioxide laser sessions
  Other Names: fractional CO2 laser
  Arms: Treatment A
Drug: Tacrolimus Oint 0.03% — topical daily tacrolimus ointment application
  Other Names: Tacrolimus Oint 0.03% (Tarolimus)

SUMMARY:
The aim the clinical trial was to find out whether fractional CO₂ laser sessions in combination with application of daily topical tacrolimus 0.03% would enhance the action of the drug and pose as a possible combination treatment option for stable vitiligo lesions. This combination treatment was applied to one side of the body and the response was compared to the response of the lesions on the other side of the body to daily topical tacrolimus 0.03% alone, which was used as control.

DETAILED DESCRIPTION:
Each patient included in the study received treatment A on the lesions on one side of his/her body, and treatment B on the other side.

Treatment A included 4 monthly sessions of fractional CO₂ laser on the lesions plus application of topical tacrolimus 0.03% (Tarolimus) on the lesions 6 hours after each session and twice daily in between the sessions and for 1 month after the last session.

Treatment B included only the application of topical tacrolimus 0.03% (Tarolimus) on the lesions twice daily for 5 months.

Fractional laser The device used was DEKA, SmartXide DOT (Dermal Optical Thermolysis), Italy fractional Carbon Dioxide Laser (fig. 8). This device is an ablative fractional 10,6000 nm CO² Laser with variable pulse duration (0.2-2 ms), 350-μm beam spot size, scanner area of 15x15 mm and penetration depth between 200 to 1,500 μm.

Tacrolimus ointment 0.03% (Tarolimus) Applied on the lesions treated by fractional CO² laser 6 hours after each laser session, then twice daily in between the sessions and 1 month after the last session.

Applied on the lesions on the other half of the body (not treated with fractional CO² laser) twice daily for 4 months.

ELIGIBILITY:
Inclusion criteria:

* Patients with stable vitiligo for at least 6 months, stability being defined as no eruption of fresh lesions and no extension of pre-existing lesions.
* Age ≧ 12 years.
* Symmetrical vitiligo.
* Three month treatment-free period.

Exclusion criteria:

* Patients younger than 12 years of age.
* Non-stable lesions.
* Non-symmetrical vitiligo.
* Patients currently on other lines of treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
repigmentation | 5 months
  reduction in Vitiligo Area Scoring Index of lesions

CONTACTS AND LOCATIONS:
Overall Officials: Ola M AbuZeid, MD, Study Director — Kasr Al Aini dermatology department; Dina ElSharkawy, MD, Study Director — Kasr Al Aini dermatology department

IPD SHARING:
Plan to Share IPD: No